CLINICAL TRIAL: NCT04102059
Title: Pattern of Work Related Musculoskeletal Disorders Among Nurses at Main Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Israa salah El-Din Shaker, principle investgator, Assiut University
Other Study IDs: WRMDsNAUH
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Work-related Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The term work-related musculoskeletal disorders (WRMDs) is defined according to the World Health Organization (WHO), as a wide range of inflammatory and degenerative diseases and disorders that result in pain and functional impairment. They arise when individuals are exposed to work activities and conditions that significantly contribute to their development or exacerbation, but which may not be their sole cause (1,2).

Another definition The National Institute for Occupational Safety and Health defined WRMDs as "an injury of the muscles, tendons, ligaments, nerves, joints, cartilage, bones, or blood vessels in the arms, legs, head, neck, or back that is caused or aggravated by work tasks such as lifting, pushing, and pulling(3-5).

They represent the second largest cause of short-term or temporary work disability after the common cold (6).Apart from lowering the quality of workers' life and reducing the productivity, WRMDs are the most expensive form of work disability, attributing to about 40% of all costs toward the treatment of work-related injuries(7).

It is estimated that almost one-third of all cases of sick leave among health care workers are related to musculoskeletal disorders(8).According to the Bureau of Labor Statistics (BLS) in 2013, WRMDs cases accounted for 33% of all worker injury and illness cases(9).

Most WRMSDs develop over time with usually, no single cause but various factors work in combination. According to the European Occupational Safety and Health Agency (EU-OSHA), the most common physical causes and organizational risk factors of musculoskeletal disorders (MSDs) include:

* Prolonged sitting or standing in the same position
* Performing the same task over and over
* Continuing work while injured
* Awkward and static postures
* Load handling, especially when bending and twisting
* Repetitive or forceful movements
* Vibration
* Insufficient work breaks(7,10-12).

DETAILED DESCRIPTION:
Nurses have to perform many physically demanding tasks such as transferring patients in and out of bed, lifting patients onto a bed, and continually maintaining bent-forward or twisted postures

Examples of WRMDs :

1. Muscle strain: Overstretching or overexertion of a muscle or tendon.
2. Tendonitis and tenosynovitis.
3. Nerve injury: Carpal tunnel syndrome.
4. Rotator cuff injuries (affects the shoulder)
5. Epicondylitis (affects the elbow)
6. Trigger finger.
7. Low back injuries (16,17). A previous cross-sectional study was conducted in a tertiary care hospital in Chennai (India)2013 among dentists, laboratory technicians, nurses, physicians, and physiotherapists of various clinical departments. It showed that irrespective of regions, musculoskeletal problems during last 12 months was reported by 56% of nurses 55% of physiotherapists, 54% of dentists, 39% of laboratory technicians and 38% of physicians. About half (50.7%) of the participants reported symptoms involving at least one part of their bodies. Among all the symptoms, low back pain (LBP) was the highest (45.7%), followed by neck pain (28.5%) and shoulder pain (23.5%), whereas hip/thigh pain (7.1%) and elbow pain (5%) was the least reported(7). A descriptive cross-sectional study was conducted among health care workers in Lahore, Pakistan, Muscle aches/ muscle strains were mostly reported among nurses (38.6%) (19).A cross sectional study was conducted among nurses working in Mansoura Children University Hospital during the period from January to May 2017. The prevalence of musculoskeletal complaints among nurses was 85.9 % .The most common sites were elbow (85.2%) followed by pelvis/ thigh (74.9%) and wrist (64.6%). Surprisingly the least site for pain was low back pain (37%)(20).

A cross sectional study is implemented on 135 female nurses in Suez Canal University Hospital and Ismailia About 113(83.7%) of the participants reported musculoskeletal symptoms(21).

ELIGIBILITY:
Inclusion Criteria:All nurses at Main Assiut University Hospital

-

Exclusion Criteria:

* Male nurses.
* pre-employment musculoskeletal disease.
* Autoimmune connective tissue disease.
* Previous musculoskeletal surgery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All female nurses at Main Assiut University Hospital.
Sampling Method: Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
study pattern of work related musculoskeletal disorders among nurses at Main Assiut University Hospital | through study completion, an average of 1 year
  Interview questionnaire
detect work related skeletal problems | through study completion, an average of 1 year
  x-ray on the affected area
detect muscular problems | through study completion, an average of 1 year
  Musculoskeletal examination
detect nerve affection | through study completion, an average of 1 year
  nerve conduction test

REFERENCES:
- [Background] SA A. Work- Related Musculoskeletal Symptoms Among Nurse Staff in Ismailia, Egypt. Egypt J Occup Med. 2018;42(1):61-78.
- [Result] Elsherbeny EE1, Elhadidy SS1 E-MRE-BA. Prevalence and Associated Factors of Musculoskeletal Complaints Among Nurses of Mansoura University Children Hospital. Egypt J Occup Med. 2018;42(2):151-66.